CLINICAL TRIAL: NCT02325908
Title: Evaluation of Body Hydration Status in Hemodialysis Patients Using Segmental Bioimpedance Analysis
Brief Title: Body Fluid Dynamics in Hemodialysis Patients, an Estimation of Dry Weight
Status: Terminated | Type: Observational
Sponsor: Renal Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RRI091-97
Record Dates: First submitted 2014-12-16; First posted 2014-12-25 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Kidney Disease
Keywords: Hemodialysis; Estimated Dry Weight
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — During every study day, 1 tube (3.5mL) will be collected before and 1 tube (3.5mL) after HD. This will be done at each study day until the subject reaches optimal hydration status. These samples will be used to assess Na+, K+, Ca++ concentrations and conductivity of the blood. We'll also measure aldosterone monthly.In case of technical issues (which may include device malfunction, transportation of samples, or scheduling of personnel), samples may be frozen temporarily. Samples may also be frozen and kept for future biochemical studies (see "Consent form for future biochemical studies").
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hemodialysis patients: Dialysis patients will have their estimated dry weight measured with calf segmental bioimpedance. Based on these measurements, their dry weight will be adjusted and the amount of fluid removed during subsequent dialysis treatments will be increased by 200-300mL. The additional fluid removal will occur during 3 consecutive hemodialysis sessions. In addition, these subjects will also use VStim during these treatments. to prevent common intradialytic symptoms by promoting vascular refilling.
- Healthy Controls: No Intervention was administered. Both groups had their hydration status measured with segmental bioimpedance The group of healthy subjects was studied in order to obtain a range of values for normal hydration status.

SUMMARY:
The purpose of this study is to learn how the amount of fluid in the body of a hemodialysis patient affects him or her. Body hydration is the amount of fluid in the human body and known to be related to blood pressure. Too much fluid can lead to high blood pressure which can cause heart problems and eventually lead to death. Bioimpedance Spectroscopy (BIS) is a method that may be used to measure body hydration. This can be applied in the whole body, arm, trunk, calf, and leg. It is a non-invasive and inexpensive method and no known risk. BIS measurements can be used to assess optimal hydration status which is defined as a patient's ideal weight after completing a dialysis treatment. The investigators hypothesize that your target weight may be better estimated by the BIS. The results of this study, in particular the continuous measurement of calf hydration which is associated with the hydration of the whole body, may provide useful information about physiologic ("healthy") body hydration. It may possibly help to improve treatment procedures for patients in the future. The Renal Research Institute plans to enroll 100 chronic hemodialysis patients and 200 healthy controls in this study.

DETAILED DESCRIPTION:
Estimation of the hydration state of chronic kidney disease (CKD) patients is an important aspect of clinical practice. Deterioration in renal function often leads to volume overload with resulting hypertension and there is no simple and accurate technique available to measure body hydration at the moment.

In hemodialysis (HD) patients, one limitation to adequate ultrafiltration necessary to achieve optimal hydration status (dry weight) is inadequate vascular refilling from the interstitial space. Blood pressure may decrease due to limitation of vascular refilling even when dry weight is far from being achieved. Therefore, an objective and accurate method to provide hydration state would be very useful for clinical practice. Whole body bioimpedance techniques have been used to measure body fluid volume for many years. However, it is difficult to accurately indicate the hydration state by body fluid volume of normal variations, and the accuracy of measurement is influenced by various body compositions. Recently, the investigators have proposed that hydration can be approached using a calf bioimpedance technique by monitoring change in resistance during HD. Since the lower limbs tend to contain more fluid than other body segments in ambulatory people due to the effect of gravity, measurement of the calf provides more accurate information about body hydration in the HD patient.

In this study, the investigators hypothesize that:

1. Since the degree of hydration is greater in the leg than in the arm and the trunk due to the effect of gravity, monitoring change in resistance in the whole or part of the leg will provide information as to whether optimal hydration status (a state in which excess extracellular fluid is absent) has been attained. The investigators postulate that a change in the slope of resistance curve (CSR) in the calf approaches zero as optimal hydration status is achieved.
2. Optimal hydration status can be approximated by comparison of two values: (1) measurement of local electrical resistivity in the interstitial compartment and (2) known range of resistivity in healthy subjects (HS). Combination of the normalized resistivity (μ) and CSR are considered as indicators of physiological optimal hydration status. Physiological optimal hydration status, as an objective index, is a major goal of hemodialysis so that the excess body water can be maximally removed according to this value. In practice this can be approached but should never be exceeded.

Because flattening of the curve should be verified by the near normal resistivity, a group of healthy subjects would have to be added to provide a normal range of resistivity at all ages and both sexes.

ELIGIBILITY:
Inclusion Criteria:

* Stable hemodialysis patients believed to be at all levels of hydration by their treating physician should be chosen.

Exclusion Criteria:

* Myocardial infarction or stroke in the preceding 6 months
* Two episodes of hypotension (systolic BP < 90 mmHg) during the 3 dialysis procedures preceding entering the treatment phase
* Grade IV CHF by NY classification
* Simultaneous participation in another clinical study except observational trials.
* Any psychological condition which could interfere with the patient's ability to comply with the study protocol.
* Pregnancy.
* Amputation of a limb.
* Pace maker, implantable pump, artificial joint.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stable hemodialysis patients believed to be at all levels of hydration by their treating physician will be chosen. 100 subjects will be chosen to include approximately 50% women in the hemodialysis program. Subjects will be selected from a wide range of ages and body mass indexes
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2008-04; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Dry weight as determined by segmental bioimpedance in comparison to baseline | 1 month

SECONDARY OUTCOMES:
Mean pre dialysis and post dialysis blood pressure in comparison to baseline | 1 month
Numbers and doses of blood pressure medications prescribed | 1 month
  If the blood pressure is improved based on better assessment of dry weight, the need for multiple blood pressure meds and dosing will be reduced.

CONTACTS AND LOCATIONS:
Overall Officials: Fansan Zhu, MD, Principal Investigator — Renal Research Institute

REFERENCES:
- [Result] Spiegel DM, Bashir K, Fisch B. Bioimpedance resistance ratios for the evaluation of dry weight in hemodialysis. Clin Nephrol. 2000 Feb;53(2):108-14. PMID 10711412
- [Result] Jaeger JQ, Mehta RL. Assessment of dry weight in hemodialysis: an overview. J Am Soc Nephrol. 1999 Feb;10(2):392-403. doi: 10.1681/ASN.V102392. PMID 10215341
- [Result] Leypoldt JK, Cheung AK. Evaluating volume status in hemodialysis patients. Adv Ren Replace Ther. 1998 Jan;5(1):64-74. doi: 10.1016/s1073-4449(98)70016-0. PMID 9477217
- [Result] Zhu F, Schneditz D, Wang E, Martin K, Morris AT, Levin NW. Validation of changes in extracellular volume measured during hemodialysis using a segmental bioimpedance technique. ASAIO J. 1998 Sep-Oct;44(5):M541-5. doi: 10.1097/00002480-199809000-00045. PMID 9804490
- [Result] Piccoli A. Identification of operational clues to dry weight prescription in hemodialysis using bioimpedance vector analysis. The Italian Hemodialysis-Bioelectrical Impedance Analysis (HD-BIA) Study Group. Kidney Int. 1998 Apr;53(4):1036-43. doi: 10.1111/j.1523-1755.1998.00843.x. PMID 9551415
- [Result] Katzarski K, Charra B, Laurent G, Lopot F, Divino-Filho JC, Nisell J, Bergstrom J. Multifrequency bioimpedance in assessment of dry weight in haemodialysis. Nephrol Dial Transplant. 1996;11 Suppl 2:20-3. doi: 10.1093/ndt/11.supp2.20. PMID 8803989
- [Result] Zhu F, Schneditz D, Levin NW. Sum of segmental bioimpedance analysis during ultrafiltration and hemodialysis reduces sensitivity to changes in body position. Kidney Int. 1999 Aug;56(2):692-9. doi: 10.1046/j.1523-1755.1999.00588.x. PMID 10432410
- [Result] Steuer RR, Germain MJ, Leypoldt JK, Cheung AK. Enhanced fluid removal guided by blood volume monitoring during chronic hemodialysis. Artif Organs. 1998 Aug;22(8):627-32. doi: 10.1046/j.1525-1594.1998.06036.x. PMID 9702312
- [Result] Lopot F, Kotyk P, Blaha J, Forejt J. Use of continuous blood volume monitoring to detect inadequately high dry weight. Int J Artif Organs. 1996 Jul;19(7):411-4. PMID 8841855
- [Result] Bogaard HJ, de Vries JP, de Vries PM. Assessment of refill and hypovolaemia by continuous surveillance of blood volume and extracellular fluid volume. Nephrol Dial Transplant. 1994;9(9):1283-7. PMID 7816290
- [Result] Leunissen KM, Kooman JP, van Kuijk W, van der Sande F, Luik AJ, van Hooff JP. Preventing haemodynamic instability in patients at risk for intra-dialytic hypotension. Nephrol Dial Transplant. 1996;11 Suppl 2:11-5. doi: 10.1093/ndt/11.supp2.11. PMID 8803987
- [Result] Kouw PM, Kooman JP, Cheriex EC, Olthof CG, de Vries PM, Leunissen KM. Assessment of postdialysis dry weight: a comparison of techniques. J Am Soc Nephrol. 1993 Jul;4(1):98-104. doi: 10.1681/ASN.V4198. PMID 8400074
- [Result] Franz M, Pohanka E, Tribl B, Woloszczuk W, Horl WH. Living on chronic hemodialysis between dryness and fluid overload. Kidney Int Suppl. 1997 Jun;59:S39-42. PMID 9185103
- [Result] Zhu F, Kuhlmann MK, Sarkar S, Kaitwatcharachai C, Khilnani R, Leonard EF, Greenwood R, Levin NW. Adjustment of dry weight in hemodialysis patients using intradialytic continuous multifrequency bioimpedance of the calf. Int J Artif Organs. 2004 Feb;27(2):104-9. doi: 10.1177/039139880402700205. PMID 15061473
- [Result] Frankel VH, McLeod KJ. Calf muscle pump stimulation as an adjunct to orthopaedic surgery. Surg Technol Int. 2005;14:297-304. PMID 16525986
- [Result] Madhavan G, Stewart JM, McLeod KJ. Effect of plantar micromechanical stimulation on cardiovascular responses to immobility. Am J Phys Med Rehabil. 2005 May;84(5):338-45. doi: 10.1097/01.phm.0000159970.81072.8b. PMID 15829780
- [Result] Madhavan G, Stewart JM, McLeod KJ. Cardiovascular systemic regulation by plantar surface stimulation. Biomed Instrum Technol. 2006 Jan-Feb;40(1):78-84. doi: 10.2345/0899-8205(2006)40[78:CSRBPS]2.0.CO;2. PMID 16544794
- [Result] Stewart JM, Karman C, Montgomery LD, McLeod KJ. Plantar vibration improves leg fluid flow in perimenopausal women. Am J Physiol Regul Integr Comp Physiol. 2005 Mar;288(3):R623-9. doi: 10.1152/ajpregu.00513.2004. Epub 2004 Oct 7. PMID 15472009